CLINICAL TRIAL: NCT03939481
Title: A Prospective Observational Cohort Study to Develop a Predictive Model of Taxane-Induced Peripheral Neuropathy in Cancer Patients
Brief Title: Treatment Effects on Development of Chemotherapy-Induced Peripheral Neuropathy in Patients With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S1714; NCI-2018-01568 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1714 (Other: SWOG); SWOG-S1714 (Other: DCP); S1714 (Other: CTEP); UG1CA189974 (NIH)
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Lung Non-Small Cell Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Stage I Lung Cancer AJCC v8; Stage I Ovarian Cancer AJCC v8; Stage IA Ovarian Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage IB Ovarian Cancer AJCC v8; Stage IC Ovarian Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage II Ovarian Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIA Ovarian Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage IIB Ovarian Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Ovarian Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (non-study chemo, questionnaire, assessments): Patients receive chemotherapy regimen per treating physician for 52 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete questionnaires at weeks 4, 8, 12, 24 and 52.
  Interventions: Drug: Chemotherapy; Other: Functional Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Chemotherapy — Given chemotherapy regimen
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Other: Functional Assessment — Functional and sensory clinician assessments
Other: Questionnaire Administration — Patient and physician reported responses

SUMMARY:
This trial studies treatment effects on development of chemotherapy-induced peripheral neuropathy in patients with cancer. Treatments for cancer can cause a problem to the nervous system (called peripheral neuropathy) that can lead to tingling or less feeling in hands and feet. Studying certain risk factors, such as age, gender, pre-existing conditions, and the type of treatment for cancer may help doctors estimate how likely patients are to develop the nerve disorder.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop and validate a clinical risk prediction model using clinical factors for the development of peripheral neuropathy in patients receiving taxane-based chemotherapy regimens.

SECONDARY OBJECTIVES:

I. To examine patient-reported outcomes (PROs) and objective measures of chemotherapy induced peripheral neuropathy (CIPN) to better define the phenotype of peripheral neuropathy in this patient population.

II. To assess the incidence of CIPN within one year in this patient population. III. To identify predictors of treatment dose reductions, delays, and discontinuations associated with CIPN symptoms in this patient population.

OTHER OBJECTIVES:

I. To collect serum and plasma samples for future testing for biomarker and mechanistic studies of CIPN.

OUTLINE:

Patients receive chemotherapy regimen per treating physician for 52 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete questionnaires at weeks 4, 8, 12, 24 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have stage I, II, or III primary non-small cell lung, primary breast, or primary ovarian cancer based on clinical or pathologic evaluation. Patients with Stage IV disease are not eligible.
* Patients must be planning to start treatment with a taxane-based chemotherapy as part of one of the study-approved taxane regimens (docetaxel chemotherapy regimens for treatment of breast or ovarian cancer, or paclitaxel chemotherapy regimen for treatment of breast, non-small cell lung, or ovarian cancer) within 14 days after registration. (Note that docetaxel or paclitaxel may be administered with a non-neurotoxic chemotherapy, such as cyclophosphamide, and/or biologic agent, such as trastuzumab, and/or carboplatin. Additionally, nab-paclitaxel may not be substituted for paclitaxel for purposes of this study.)
* Patients who will receive treatment in the setting of any other clinical trial are eligible as long as it is one of the study-approved regimens. Patients may receive additional treatments (i.e., experimental therapy, immunotherapy, biologics, etc.) as part of another clinical trial in addition to any regimen approved in this study.
* Patients must not have received a taxane (paclitaxel, docetaxel, or protein-bound paclitaxel), platinum (cisplatin, carboplatin, or oxaliplatin), vinca alkaloid (vinblastine, vincristine, or vinorelbine), or bortezomib-based chemotherapy regimen prior to registration. (Note that while patients must not have received carboplatin in the past, patients may receive a carboplatin-containing regimen after registration as part of the docetaxel or paclitaxel regimen.)
* Patients who can complete Patient-Reported Outcome (PRO) instruments in English or Spanish must:

  * Agree to complete PROs at all scheduled assessments
  * Complete the baseline PRO forms prior to registration
* Patients with pre-existing neuropathy are eligible, including those with diabetes and neurological conditions such as multiple sclerosis or Parkinson?s disease.
* Patients must agree to submit required specimens for defined translational medicine.
* Patients must be offered the opportunity to submit additional optional specimens for future, unspecified translational medicine and banking. With patient?s consent, specimens must be submitted.
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with stage I, II, or III primary non-small cell lung, primary breast, or primary ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 1336 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Development of peripheral neuropathy | Up to 24 weeks
  Will be measured as an absolute increase of >= 8 points over the baseline chemotherapy-induced peripheral neuropathy (CIPN)-20 sensory neuropathy subscale score. Will be collected before or at the 24-week assessment as the taxane-based chemotherapy regimens in this study are expected to be completed within 8 to 18 weeks. The presence of CIPN will be captured at 52 weeks to evaluate the duration of neuropathy which is anticipated to wane after treatment discontinuation.

SECONDARY OUTCOMES:
CIPN symptoms | Up to 52 weeks
  Patients experiencing a treatment change attributed to CIPN symptoms
Dose Changes | Up to 52 weeks
  Dose reductions, delays, and discontinuations of treatment (prior to completing the original treatment plan)
Health-related Quality of Life | Up to 52 weeks
  Assessed using the Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29). The PROMIS-29 is a well validated assessment tool that offers both qualitative and quantitative measures of health-related quality of life. The PROMIS-29 includes 29 questions evaluating areas of physical function, anxiety, depression, fatigue, sleep, social functioning, and pain interference. The PROMIS-29 assesses severity levels of symptoms and their effect on the patient's functioning.
Visual Analog Toxicity Score | Up to 52 weeks
  Assessed using the Visual Analog Toxicity Score. The Visual Analog Toxicity Score is a single question asking the physician to rate how the physician feels the patient's disease and treatment affects their daily life on a scale from 0 (no symptoms and no effect on life) to 10 (severe effects of treatment and patient would rather be dead).
Patient Reported Symptom | Up to 52 weeks
  Assessed using the Patient Reported Symptom Burden Score. The Patient Reported Symptom Score at baseline contains one question to assess how cancer symptoms affect the patient's life (scale 0 [no burden at all] to 10 [a great burden]). At follow-up, the Symptom Burden Score contains five questions: 1) to assess burden of side effects of cancer treatment on life (scale 0 [no burden at all] to 10 [a great burden]), 2) to assess severity of side effects from cancer treatment (scale 0 [no side effects]) to 10 [side effects extremely severe and unbearable]), 3) to assess tolerability of side effects for set time periods (yes/no), 4) to assess level at which treatment would be considered intolerable (scale 0 [side effects not severe at all] to 10 [side effects extremely severe and unbearable]), and 5) to assess the burden of cancer symptoms and treatment symptoms (scale 0 [no burden at all] to 10 [a great burden]).
Leisure-time Exercise Habits | Up to 52 weeks
  Assessed using the Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ). The GSLTPAQ is a brief 4 item self-administered questionnaire of usual leisure-time exercise habits over a typical 7-day period. The Leisure Score Index (LSI) is calculated based on the first 3 questions. The LSI scores can be used to classify respondents into active (LSI > 24) and insufficiently active (LSI < 23) categories.
Patient-Reported Outcomes | Up to 52 weeks
  Assessed using the Patient Reported Outcomes Common Terminology Criteria for Adverse Events (PRO-CTCAE [CTCAE Version 5.0]). PRO-CTCAE assesses 78 adverse events by self-report with 124 items. Each item uses a plain language term for the adverse event, the attribute of interest, and the standard recall period of "the past 7 days".
National Cancer Institute-Common Terminology Criteria for Adverse Events | Up to 52 weeks
  The NCI-CTCAE is a subjective method to evaluate CIPN performed by a healthcare professional. The treating physician will grade the subject's dysesthesia, paresthesia, neuralgia, peripheral sensory neuropathy, and peripheral motor neuropathy on a scale of 0 to 5 depending on the severity. The advantage of the NCI-CTCAE is that the assessment is quick and easy for providers to perform, (8) but it is limited by the subjectivity of interpretation, lack of detail about location, type, and severity of impairment, and narrow scoring range.
Assess incidence of CIPN | Up to 52 weeks
  Assessed using European Organization for Research and Treatment of Cancer (EORTC) QLQ-CIPN20 (CIPN-20). The EORTC QLQ-CIPN20 is a 20-item questionnaire that evaluates CIPN using 3 subscales that assess sensory (9 items), motor (8 items), and autonomic (3 items) symptoms and functioning with each item measured on a 1-4 scale (1, not at all; 4, very much). The sensory subscale raw scores range from 1 to 36. The CIPN-20 subscale raw scores are linearly converted to a 0-100 scale such that a high score corresponds to a worse condition or more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Meghna S Trivedi, Principal Investigator — SWOG Cancer Research Network
Locations (169):
- United States (166):
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Little Company of Mary Hospital, Evergreen Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Saint Joseph Hospital, Nashua, New Hampshire
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Randolph Hospital, Asheboro, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Nash General Hospital, Rocky Mount, North Carolina
  - NHRMC Radiation Oncology - Supply, Supply, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Kaiser Permanente Northwest, Portland, Oregon
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - Kent Hospital, Warwick, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
- Instituto Nacional del Cancer, Independence, Chile
- Instituto Nacional De Cancerologia, Bogotá, Colombia
- Instituto Nacional De Cancerologia de Mexico, Mexico City, Tlalpan, Mexico